CLINICAL TRIAL: NCT04397497
Title: A Randomized, Double Blind, Placebo-controlled Trial of Mavrilimumab for Acute Respiratory Failure Due to COVID-19 Pneumonia With Hyper-inflammation (the COMBAT-19 Trial)
Brief Title: Mavrilimumab in Severe COVID-19 Pneumonia and Hyper-inflammation (COMBAT-19)
Acronym: COMBAT-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Lorenzo Dagna, Head, Unit of Immunology Rheumatology Allergy and Rare Diseases (UnIRAR), Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COMBAT-19
Record Dates: First submitted 2020-05-20; First posted 2020-05-21 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Covid-19; Acute Respiratory Failure; ARDS, Human; Sars-CoV2; Viral Pneumonia
Keywords: covid-19; Acute respiratory failure; mavrilimumab; GM-CSF; GM-CSF receptor alpha; SARS-CoV2; viral pneumonia
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome; Pneumonia, Viral | interventions — mavrilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mavrilimumab (Experimental): Single dose of IV Mavrilimumab
  Interventions: Drug: Mavrilimumab
- Placebo (Placebo Comparator): Single dose of matching IV placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mavrilimumab — human monoclonal antibody targeting GM-CSF receptor-alpha
  Other Names: KPL-301; CAM-3001
  Arms: Mavrilimumab
Drug: Placebo — matching volume of diluent
  Arms: Placebo

SUMMARY:
This study is a prospective, phase II, multi-center, randomized, double-blind, placebo-controlled trial to evaluate the efficacy and safety of mavrilimumab in hospitalized patients with acute respiratory failure requiring oxygen supplementation in COVID- 19 pneumonia and a hyper-inflammatory status. The study will randomize patients to mavrilimumab or placebo, in addition to standard of care per local practice. The total trial duration will be 12 weeks after single mavrilimumab or placebo dose.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of mavrilimumab versus placebo in addition to best standard of care (SoC) in the treatment of COVID-19 pneumonia.

As of May 13, 2020, COVID-19 has been confirmed in more than 4.2 million people worldwide. Mortality rate has been reported to be approximately 3.7%, which is nearly 4 times higher than that of influenza: there is an urgent need for effective treatment.

Accumulating evidence suggests that patients with severe acute COVID-19 pneumonia have a cytokine storm syndrome, or unbalanced hyper-inflammatory response resulting in markedly elevated cytokine and chemokine production.

GM-CSF is a cytokine with dual roles as a critical pulmonary hormone and proinflammatory properties that can exaggerate tissue inflammation. Recent preliminary uncontrolled clinical observations on 13 non-mechanically-ventilated patients in the promoter institution suggest that GM-CSF pathway blockade with mavrilimumab is an effective and well-tolerated treatment for COVID-19 pneumonia.

We will perform a prospective, phase II, multi-center, randomized, double-blind, placebo-controlled trial to evaluate the efficacy and safety of mavrilimumab in hospitalized patients with acute respiratory failure requiring oxygen supplementation in COVID- 19 pneumonia and a hyper-inflammatory status. The study will randomize non-mechanically-ventilated adult patients to mavrilimumab or placebo, in addition to standard of care per local practice, which may include but not limited to anti-viral treatment, hydroxychloroquine, low-dose corticosteroids (≤ 10 mg of prednisone or equivalent) and/or supportive care. The total trial duration will be 12 weeks after single mavrilimumab or placebo infusion. Safety will be closely monitored by a dedicated external data safety monitoring board (DSMB) at regular intervals during the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years of age)
* Signed informed consent by any patient capable of giving consent, or, when the patient is not capable of giving consent, by his or her legal/authorized representative or according to local guidelines
* Patients clinically diagnosed with SARS-CoV-2 virus by PCR or by other approved diagnostic methodology
* Hospitalized with COVID-19-induced pneumonia evidenced by chest x-ray or CT scan with pulmonary infiltrates
* Patient requiring oxygen supplementation (i.e. with a SpO2 ≤ 92% while breathing room air) and having a PAO2/FIO2 ratio ≤ 300 mmHg
* Lactate dehydrogenase (LDH) > normal range and at least one of the following:

  1. fever > 38.0 °C;
  2. increased levels of C-reactive Protein (CRP) ≥ 10x UNL mg/L (≥ 60 mg/l);
  3. increased levels of ferritin ≥ 2.5x UNL ( ≥ 1000 μg/L)

Exclusion Criteria:

* Onset of COVID-19 pneumonia symptoms (i.e. dyspnea/respiratory insufficiency) >14 days
* On mechanical ventilation at the time of randomization
* A PaO2/FiO2 < 100 mmHg
* Uncontrolled systemic infection (other than COVID-19)
* Hypersensitivity to the active substance or to any of the excipients of the experimental drug
* Total neutrophil count < 1500/mm3
* Severe hepatic cirrhosis
* History of chronic HBV or HCV infection
* Known or active tuberculosis (TB) or a history of incompletely treated TB; suspected or known extrapulmonary tuberculosis
* Moderate/severe heart failure (NYHA Class 3 or 4)
* Any prior (within the defined periods below) or concurrent use of immunosuppressive therapies including but not limited to the following:

  1. Anti-IL-6, anti-IL-6R antagonists or Janus kinase inhibitors (JAKi) in the past 30 days or plans to receive during the study period;
  2. Cell-depleting agents (e.g., anti CD20) without evidence of recovery of B cells to baseline level;
  3. Anakinra within 1 week of baseline; canakinumab within 8 weeks of baseline; abatacept within 8 weeks of baseline.
  4. Tumor necrosis factor (TNF) inhibitors within 2-8 weeks (etanercept within 2 weeks, infliximab, certolizumab, golimumab, or adalimumab within 8 weeks), or after at least 5 half-lives have elapsed, whichever is longer;
  5. Alkylating agents including cyclophosphamide (CYC) within 6 months of baseline;
  6. Cyclosporine (CsA), azathioprine (AZA) or mycophenolate mofetil (MMF) or leflunomide or methotrexate within 4 weeks of baseline.
* Pregnancy or lactation (Note: Women of childbearing age should use effective contraception/abstinence after treatment with mavrilimumab and for 3 months after the dosing)
* Any serious medical condition or abnormality of clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
* In the opinion of the investigator, progression to death is imminent and highly likely within the next 24 hours, irrespective of the provision of treatments
* Current participation in any other interventional investigational trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-05-22 (Estimated); Primary Completion 2020-09-22 (Estimated); Study Completion 2020-11-22 (Estimated)

PRIMARY OUTCOMES:
Reduction in the dependency on oxygen supplementation | within day 14 of treatment
  Time to the absence of need for oxygen supplementation (time to first period of 24 hrs with a SpO2 of 94%) within day 14 of treatment, stated as Kaplan- Mayer estimates of the proportion of patients on room air at day 14 and median time to room air attainment in each arm

SECONDARY OUTCOMES:
Proportion of responders (using the WHO 7-point ordinal scale) | Day 7, 14, and 28
  Response is defined as a 7-point ordinal scale of 3 or less, i.e. no supplemental oxygen
Time to response (using the WHO 7-point ordinal scale) | Within day 28 of intervention
  Time from date of randomization to the date with a 7-point ordinal scale of 3 or less, i.e. no supplemental oxygen
Proportion of improving patients (using the WHO 7-point ordinal scale) | At day 7, 14, and 28
  Proportion of patients with at least two-point improvement in clinical status
Time to resolution of fever | Within day 28 of intervention
  Time to resolution of fever (for at least 48 hours) in absence of antipyretics, or discharge, whichever is sooner
Reduction in case fatality | Within day 28 of intervention
  COVID-19-related death
Proportion of patient requiring mechanical ventilation/deaths | Within day 14 of intervention
  Proportion of hospitalized patients who died or required mechanical ventilation (WHO Categories 6 or 7)
Change in biochemical markers | Within day 28 of intervention or discharge -whatever comes first
  Change of the following serological markers over follow-up (C-reactive protein; Ferritin; D-Dimer)
Median changes in the National Early Warning Score 2 (NEWS2) | At day 7, 14, and 28
  Median changes of NEWS2 score from baseline
Time to clinical improvement as evaluated with the National Early Warning Score 2 (NEWS2) | Within day 28 of intervention or discharge -whatever comes first
  Time to clinical improvement (as defined as a NEWS2 score of 2 or less maintained for at least 24 hours or discharge, whichever comes first)
Variations in radiological findings | Within day 28 of intervention or discharge -whatever comes first
  Variations from baseline to subsequent timepoints (when available) in terms of percentage of lung involvement, modifications in the normal parenchyma, ground glass opacities (GGO), crazy paving pattern,parenchymal consolidations, and evolution towards fibrosis.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | By day 84
  Number of patients with treatment- related side effects (as assessed by Common Terminology Criteria for Adverse Event (CTCAE) v.5.0), serious adverse events, adverse events of special interest, clinically significant changes in laboratory measurements and vital signs

OTHER OUTCOMES:
Clinical efficacy of mavrilimumab compared to the control arm by clinical severity | Within day 28 of intervention
  To evaluate the primary and secondary endpoints in different subgroups of patients:
  * mild respiratory failure: PaO2/FiO2 ≤ 300 and > 200 mmHg;
  * moderate respiratory failure: PaO2/FiO2 ≤ 200 and > 100 mmHg
Changes in serum IL-6 (exploratory biomarker) | By day 84
  Median changes in serum IL-6
Changes in serum IL-1RA (exploratory biomarker) | By day 84
  Median changes in serum IL-1 receptor antagonist
Changes in serum TNF-alpha (exploratory biomarker) | By day 84
  Median changes in serum TNF-alpha
Changes in CBC + differential (exploratory biomarker) | By day 84
  Median variations in haemoglobin and leucocyte counts
Level of anti-SARS-CoV2 antibodies (exploratory biomarker) | By day 84
  Median titres od anti-SARS-CoV2 antibodies
Virus eradication (exploratory biomarker) | By day 84
  Proportion of patients with a positive swab for SARS-CoV2 by PCR
Anti-drug antibodies (exploratory biomarker) | By day 84
  Proportion of patients who developed anti-drug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Dagna, MD, Principal Investigator — Ospedale San Raffaele
Locations (3):
- Italy (3):
  - IRCCS Policlinico San Donato, San Donato, MI
  - IRCCS Ospedale San Raffaele, Milan
  - IRCCS Istituto Ortopedico Galeazzi, Milan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR